CLINICAL TRIAL: NCT06472596
Title: Risk of Developing Chronic Kidney Disease in Patients With Bronchial Asthma at Sohag University Hospitals
Brief Title: Risk of Chronic Kidney Disease in Bronchial Asthma
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marihan Nazmy Shehata, doctor resident at pediatric department in sohag university hospitals, Sohag University
Other Study IDs: soh-Med-24-05-11MS
Record Dates: First submitted 2024-06-10; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma | interventions — Blood Cell Count; Blood Gas Analysis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cases ( asthmatic patients): asthmatics investigated by serum creatinine , GFR calculation , ESR,CRP,ABG,CBC , serum electrolytes , interleukin6, tumor necrotic factor alpha
  Interventions: Diagnostic Test: CBC, CRP ,ESR, ABG , interleukin 6, tumor necrotic factor alpha
- control (healthy persons): healthy persons investigated by same investigations and compare results with asthmatics
  Interventions: Diagnostic Test: CBC, CRP ,ESR, ABG , interleukin 6, tumor necrotic factor alpha

INTERVENTIONS:
Diagnostic Test: CBC, CRP ,ESR, ABG , interleukin 6, tumor necrotic factor alpha — compare results of investigations in asthmatics and non asthmatics

SUMMARY:
the study aims to determine the frequency and factors associated with chronic kidney disease among asthmatic patients in order to determine persons who are at risk of developing chronic kidney disease and require strict follow up in long run , to evaluate severity of asthma as a potential risk for developing kidney injury , to evaluate relationship between different inflammatory markers with severity of asthma and risk of deneloping chronic kidney disease

ELIGIBILITY:
Inclusion Criteria:

* all children diagnosed as bronchial asthma at sohag university hospitals from age of 2 years to age of 18 years and donot have any associated disease

Exclusion Criteria:

* persons who have any chronic illness persons who have any associated disease with bronchial asthma persons who missing clinical and laboratory investigations persons who refusing to give written informed consent for the study

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: cases (asthmatics) and control ( healthy ) from age of 2 years to 18 years
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-11 (Estimated)

PRIMARY OUTCOMES:
change in kidney function in asthmatics | change in kidney function in asthmatics after diagnosis and start treatment through out the duration of study (an average 1 year )
  change in serum creatinine , GFR calculation

CONTACTS AND LOCATIONS:
Locations (1):
- Marihan Nazmy Shehata, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No